CLINICAL TRIAL: NCT00808431
Title: ST of TN-Salud Con La Familia: Prevent Onset of Ped Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Shari Barkin, MD, MSHS, Professor of Pediatrics, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 080673
Record Dates: First submitted 2008-12-04; First posted 2008-12-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Obesity
Keywords: Obesity; Diabetes; Physical Activity; Child Feeding; Growth Trajectories; Family based
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): Lifestyle counseling
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — 3 month skills building program emphasizing parent training, behavior modification training, nutrition education, and physical activity promotion
  Other Names: Salud con la familia

SUMMARY:
Preventing the onset of pediatric obesity and diabetes in Latino families

The investigators will conduct a randomized controlled trial of a family-based community centered intervention. One-hundred Latino families with children ages 3-5 will be randomly allocated to either the intervention group (a 3-month skills building program to improve nutrition and aerobic activity for child-parent dyads) or a control group (literacy promotion). Through an active partnership with Nashville Metro Parks and Recreation and the Division of General Pediatrics at the Vanderbilt Children's Hospital, the investigators will: 1) Implement an intervention for Latino families with young children that includes parent training, behavior modification training, nutrition education, and physical activity promotion; 2) Evaluate how this intervention affects growth trajectories in children; 3) Evaluate how this intervention affects parenting practices for Latino families to improve nutrition and physical activity; and 4) Evaluate the ability to link families into a pediatric medical home if they have none identified. By developing innovative family-focused interventions, finding solutions to health conditions such as obesity and diabetes could be realized-con la familia.

DETAILED DESCRIPTION:
Obesity is a well-known risk factor for the development of diabetes. Obesity rates have rapidly increased over the past three decades for all Americans and have doubled for children. Latino children experience obesity at disproportionate rates. The most promising obesity interventions have focused on having children partner with a parent to set goals. Latino cultural norms emphasizing family provide a unique opportunity to develop family-centered interventions.

We will recruit 100 families (child-parent dyad) via a multi-pronged strategy including: provision of bilingual informational flyers; announcements on a Spanish radio program; and additional strategies developed by key community leaders in the Nolensville corridor. This recruitment approach has been successful for us in the past. Once recruited into the program, parent-child dyads will be randomly allocated to either the intervention group or control group (described below).

Intervention Group

Fifty (50) families will be randomly allocated to receive the Salud Con La Familia skills building curriculum at Coleman Community Center, which will include:

1. Twelve (12) weekly 60-minute sessions in the recreation center (Refer to Table 1). The parent-child dyad will participate in 4 sessions from the En Sus Marcas curriculum, which was just tested by this study team (Barkin, PI). These sessions emphasize skills building around parenting, behavior modification, daily physical activity, and decreased sedentary activity. To this we will add 8 sessions from the Salud, Salsa, y Sabor25 curriculum, a best-practice program to improve nutrition and energy balance for Latino families, designed by the National Latino Children's Institute (NLCI) but not yet utilized in Tennessee. The combination of these two promising curricula results in a comprehensive program that includes all ADA-recommended elements of effective interventions for pediatric overweight.23 All sessions will be led by the same bilingual facilitators to ensure maximum fidelity and minimal difference between the information provided to participants. While this program has been designed in active partnership with Nashville Metro Parks and Recreation, we are also currently conducting a listening tour with key informants from the Nolensville community to provide further input into the content and implementation of the Salud Con La Familia approach. Throughout, emphasis is placed on healthy lifestyles, not on weight loss or obesity.
2. At the end of each session, the study team will facilitate creating a parent-child contract to develop concrete weekly goals around nutrition and physical activity. Such contracts are integral to behavior modification.26
3. The study team will assess if families have an identified pediatric medical home and use this for preventive health visits. If no medical home is identified, the team will assist with this health connection.

Control Group Fifty (50) families will be allocated to participate monthly with a literacy promotion skills-building curriculum. They will receive flyers when family events are offered at the community center. They will participate in data collection at the same time-points as the intervention families. Refer to Table 2 for our project timeline.

Outcomes will include: growth trajectories, parenting practices, activity patterns, and link to medical home.

ELIGIBILITY:
Inclusion Criteria:

* Latino parents with children ages 3-5
* parent agrees to participate in all sessions
* parent can be reached via telephone contact over next 3 months

Exclusion Criteria:

* non-Latino parents
* children outside target age range
* parent not agreeing to participate in all sessions
* parent cannot be reached via telephone contact over next 3 months

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Growth trajectories (using BMI, waist circumference), body composition | 3 months

SECONDARY OUTCOMES:
Physical activity accelerometry change over time, parental self-efficacy, child feeding questionnaire (parental food habits), identification of medical home | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shari Barkin, MD, MSHS, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Coleman Community Recreation Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Barkin SL, Gesell SB, Po'e EK, Escarfuller J, Tempesti T. Culturally tailored, family-centered, behavioral obesity intervention for Latino-American preschool-aged children. Pediatrics. 2012 Sep;130(3):445-56. doi: 10.1542/peds.2011-3762. Epub 2012 Aug 6. PMID 22869834